CLINICAL TRIAL: NCT05937997
Title: Evaluation and Timing in an ERAS-like Structured Rehabilitation Program After Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Median (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Johannes Schroeter, Dr. med. Johannes Schroeter, Median
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WS2017
Record Dates: First submitted 2023-06-06; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Pain Syndrome
Keywords: Enhanced recovery after surgery; spinal injuries; rehabilitation; recurrence; low back pain
MeSH Terms: conditions — Somatoform Disorders; Spinal Injuries; Recurrence; Low Back Pain

STUDY DESIGN:
Intervention Model Description: 3 therapy groups receiving different intensity of training
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A high intensity (Active Comparator): Physiotherapy with high intensity and no restrictions
  Interventions: Procedure: high intensity physiotherapy
- Group B moderate intensity (Active Comparator): Physiotherapy with medium intensity and some restrictions
  Interventions: Procedure: moderate intensity physiotherapy
- Group C low intensity (Active Comparator): Physiotherapy with low intensity and many restrictions
  Interventions: Procedure: low intensity physiotherapy

INTERVENTIONS:
Procedure: high intensity physiotherapy — high intensity exercises for 3 weeks inpatient rehabilitation
  Arms: Group A high intensity
Procedure: moderate intensity physiotherapy — moderate intensity exercises for 3 weeks inpatient rehabilitation
  Arms: Group B moderate intensity
Procedure: low intensity physiotherapy — low intensity exercises for 3 weeks inpatient rehabilitation
  Arms: Group C low intensity

SUMMARY:
The goal of this clinical trial is to investigate the safety of early inpatient rehabilitation after lumbar spine surgery.

Participants are assigned to therapy groups C (low) - A (high) intensity and receive standardized multimodal rehabilitation for 3 weeks. Groups are compared in terms of safety, disability impairment as well as pain. Timing of rehabilitation is considered.

DETAILED DESCRIPTION:
Purpose Literature on early rehabilitation after lumbar spine surgery trends towards a structurized program beginning in the post-acute phase, but publications are rare. Therefore, this study was conducted to investigate the safety of early rehabilitation according to ERAS® principles after different lumbar spine surgeries with regard to training intensity and timing of rehabilitation.

Methods Study design was prospective, non-randomized, and multicentric (3 inpatient rehabilitation facilities in Germany). Based on the senior rehabilitation physician's assessment for patient's physical capacity, patients were assigned to therapy groups C - A (low - high intensity). For statistical analysis patients were also grouped in 3 different time intervals depending on days past surgery until rehabilitation start and. Safety (recurrence rates), disability (Oswestry Disability Index (ODI)), and pain (Visual Analogue Scale (VAS)), were measured at the beginning and at the end of rehabilitation stay. Scores were compared between 3 therapy groups and 3 time intervals for within- and between-group differences. Analgesics and back orthesis use was assessed and analysed as well.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to inpatient rehabilitation facility after lumbar spine surgery

Exclusion Criteria:

* non-German speakers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Change of Oswestry Disability Index | at admission to rehabilitation clinic and at about 3 weeks at discharge
  Questionnaire with 10 items to evaluate the disability from back pain, results presented in precentage with 0 % experiencing no disability because of back issues and with 100 % experiencing the most disability because of back issues

SECONDARY OUTCOMES:
Change of Visual Analogue Scale | at admission to rehabilitation clinic and at about 3 weeks at discharge
  Standardized tool to measure subjective pain with 0 points meaning no pain and 10 points meaning the most imaginable pain
Recurrence rate | at admission to rehabilitation clinic and at about 3 weeks at discharge
  Recurrence rate of lumbar spine injuries happening throughout the interventional phase

CONTACTS AND LOCATIONS:
Locations (1):
- MEDIAN Clinics, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: Undecided
data available on reasonable request

REFERENCES:
- [Result] Schroter J, Lechterbeck M, Hartmann F, Gercek E. [Structured rehabilitation after lumbar spine surgery : subacute treatment phase]. Orthopade. 2014 Dec;43(12):1089-95. doi: 10.1007/s00132-014-3051-2. German. PMID 25413281